CLINICAL TRIAL: NCT01395758
Title: A Phase 2 Randomized Open-label Study of Erlotinib Plus Tivantinib (ARQ 197) Versus Single Agent Chemotherapy in Previously Treated KRAS Mutation Positive Subjects With Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: Erlotinib Plus Tivantinib (ARQ 197) Versus Single Agent Chemotherapy in Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ArQule, Inc., a subsidiary of Merck Sharp & Dohme LLC, a subsidiary of Merck & Co., Inc. (Rahway, NJ USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARQ 197-218
Record Dates: First submitted 2011-07-01; First posted 2011-07-18 (Estimated); Results first posted 2018-04-03 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Metastatic Non-Small Cell Lung Cancer
Keywords: KRAS mutation; metastatic NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — ARQ 197; Erlotinib Hydrochloride; Pemetrexed; Docetaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- tivantinib (ARQ 197) plus erlotinib arm (Experimental): Eligible subjects will be randomly assigned to receive erlotinib plus tivantinib (ARQ 197).
  Treatment will be open-label and continue until progression of disease, unacceptable toxicity, or another discontinuation criterion is met.
  Interventions: Drug: ARQ 197 plus erlotinib
- Chemotherapy arm (Active Comparator): Investigator's choice of single agent chemotherapy (pemetrexed, docetaxel, or gemcitabine) administered in 3-week cycles according to the approved label until disease progression or unacceptable toxicity. Subjects who discontinued chemotherapy can be switched to the crossover arm (tivantinib plus erlotinib) and continue treatment until disease progression or unacceptable toxicity.
  Interventions: Drug: Pemetrexed, docetaxel or gemcitabine

INTERVENTIONS:
Drug: ARQ 197 plus erlotinib — Eligible subjects will be randomly assigned to receive erlotinib plus ARQ 197.
  Other Names: Tivantinib
  Arms: tivantinib (ARQ 197) plus erlotinib arm
Drug: Pemetrexed, docetaxel or gemcitabine — Investigator's choice of a single agent chemotherapy (pemetrexed, docetaxel, or gemcitabine) administered according to the approved label.
  Arms: Chemotherapy arm

SUMMARY:
The purpose of this study is to evaluate progression-free survival among subjects with KRAS mutation positive Non-Small Cell Lung Cancer (NSCLC) treated with erlotinib plus tivantinib (ARQ 197) compared to single agent chemotherapy.

DETAILED DESCRIPTION:
This is a randomized, open-label Phase 2 study designed to compare treatment with erlotinib plus tivantinib (ARQ 197) versus single agent chemotherapy in subjects with previously treated KRAS mutation positive NSCLC. Eligible subjects are randomly assigned to receive erlotinib plus tivantinib or one of three (based on Investigator's choice) single-agent chemotherapy agents including pemetrexed, docetaxel, or gemcitabine.

ELIGIBILITY:
Inclusion Criteria:

1. Provide signed and dated informed consent prior to study-specific screening procedures
2. Male or female at least 18 years of age
3. Histologically or cytologically confirmed inoperable locally advanced or metastatic (stage IVA/IVB) NSCLC
4. Documented KRAS mutation positive status (per Lung Cancer Mutation Consortium [LCMC] guidelines; see www.golcmc.com)
5. At least one prior chemotherapy regimen for advanced NSCLC
6. Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria, Version 1.1
7. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
8. Male or female subjects of child-producing potential must agree to use double barrier contraception, oral contraceptives or avoidance of pregnancy measures during the study and for 90 days after the last day of treatment
9. Females of childbearing potential must have a negative serum pregnancy test
10. Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 × upper limit of normal (ULN) or ≤ 5 × ULN with metastatic liver disease
11. Total bilirubin ≤ 1.5 × ULN
12. Serum creatinine ≤ 1.5 × ULN
13. Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
14. Platelets ≥ 100 x 10^9/L
15. Hemoglobin ≥ 10 g/dL (transfusion is allowed at least 7 days prior to randomization)
16. Subjects must agree to allow testing for c-Met status if archival and/or fresh tissue biopsy samples are available.

Exclusion Criteria:

1. Previous receipt of erlotinib or other epidermal growth factor receptor (EGFR) inhibitors
2. Previous receipt of any c-MET inhibitor (a receptor tyrosine kinase) or other c-MET-targeted therapy, including ARQ 197, MetMab, crizotinib
3. Prior receipt of chemotherapy agent selected for administration in this study (e.g., if subject was treated with gemcitabine, he is not eligible to receive gemcitabine in this study but eligible to receive pemetrexed or docetaxel).
4. Inability or unwillingness to receive ARQ 197, erlotinib, docetaxel, gemcitabine, and/or pemetrexed including contraindications, hypersensitivity, or prior administration
5. Receipt of any anti-tumor treatment for NSCLC within 3 weeks (2 weeks for radiotherapy) prior to randomization
6. Pregnant or breastfeeding
7. Significant gastrointestinal disorder that could, in the opinion of the Investigator, interfere with the absorption of ARQ 197 and/or erlotinib
8. Any other significant co-morbid conditions that in the opinion of the Investigator would impair study participation or cooperation
9. Other malignancies within the last three years, with the exception of adequately treated intraepithelial carcinoma of the cervix uteri, prostate carcinoma with a prostate-specific antigen (PSA) value < 0.2 ng/mL or basal or squamous cell carcinoma of the skin
10. Known human immunodeficiency virus (HIV), or active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
11. Major surgical procedure within 4 weeks prior to randomization
12. History of cardiac disease: Congestive heart failure defined as Class II to IV per New York Heart Association classification; Active coronary artery disease; Previously diagnosed bradycardia or other cardiac arrhythmia defined as ≥ Grade 2 according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.0, or uncontrolled hypertension; Myocardial infarction that occurred within 6 months prior to study entry (myocardial infarction that occurred > 6 months prior to study entry is permitted)
13. Clinically unstable central nervous system metastasis (to be enrolled in the study, subjects must have confirmation of stable disease by MRI or CT scan within 4 weeks of randomization and have central nervous system [CNS] metastases well controlled by steroids, anti-epileptics or other symptom-relieving medications)
14. Known EGFR-mutation positive status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2011-07; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Stanford, California
  - Washington D.C., District of Columbia
  - Weston, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Kansas City, Kansas
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Burlington, Massachusetts
  - New York, New York
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Tivantinib Plus Erlotinib Arm: Tivantinib 360 mg twice daily (BID) (total daily dose 720 mg) plus erlotinib 150 mg once daily (QD), tablets, orally in 3-week cycles until disease progression or unacceptable toxicity
- Chemotherapy Arm: Investigator's choice of single agent chemotherapy (pemetrexed, docetaxel, or gemcitabine) administered in 3-week cycles according to the approved label until disease progression or unacceptable toxicity. Subjects who discontinued chemotherapy could be switched to the Crossover Arm (tivantinib plus erlotinib) and continue treatment until disease progression or unacceptable toxicity.
- Crossover Arm: Following radiographically confirmed progression, subjects in the Chemotherapy Arm had the option to enroll in the Crossover Arm to receive tivantinib plus erlotinib.
  Crossover subjects were treated with tivantinib 360 mg BID (total daily dose 720 mg) plus erlotinib 150 mg QD, tablets, orally in 3-week cycles until disease progression or unacceptable toxicity.
Period: Open-label Treatment Period
Arm/Group | Tivantinib Plus Erlotinib Arm | Chemotherapy Arm | Crossover Arm
Started | 51 | 45 | 0
Completed | 47 | 45 | 0
Not Completed | 4 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 0
Period: Crossover Period
Arm/Group | Tivantinib Plus Erlotinib Arm | Chemotherapy Arm | Crossover Arm
Started | 0 | 0 | 26
Completed | 0 | 0 | 26
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Tivantinib Plus Erlotinib Arm: Tivantinib 360 mg BID (total daily dose 720 mg) plus erlotinib 150 mg QD, tablets, orally in 3-week cycles until disease progression or unacceptable toxicity
- Total: Total of all reporting groups
Arm/Group | Tivantinib Plus Erlotinib Arm | Chemotherapy Arm | Total
Number analyzed (Participants) | 51 | 45 | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 16 | 44
  >=65 years | 23 | 29 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (9.23) | 65.2 (9.55) | 63.8 (9.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 30 | 63
  Male | 18 | 15 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 50 | 45 | 95
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 47 | 41 | 88
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 51 | 45 | 96
Cigarette Use [Count of Participants; unit: Participants]
  Yes | 46 | 42 | 88
  No | 5 | 3 | 8
Weight [Mean (Standard Deviation); unit: kilograms] | 72.50 (17.31) | 68.86 (15.19) | 70.79 (16.37)
Height [Mean (Standard Deviation); unit: centimeters] | 166.38 (10.28) | 164.88 (9.42) | 165.68 (9.86)
Eastern Cooperative Oncology Group (ECOG) Performance Status Score [Count of Participants; unit: Participants] — Grade 0: Normal activity, fully active. Able to carry on all pre-disease performance without restriction.
  Grade 1: Symptoms, but ambulatory. Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature (e.g., light housework, office work) Grade 2: In bed < 50% of the time. Ambulatory and capable of all self-care, but unable to carry out work activities. Up and about more than 50% of waking hours.
  Participants
    Grade 0 | 12 | 8 | 20
    Grade 1 | 32 | 33 | 65
    Grade 2 | 7 | 4 | 11
Confirmation of Kirsten rat sarcoma (KRAS) Mutation [Count of Participants; unit: Participants]
  Yes | 51 | 45 | 96
  No | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Among Subjects With KRAS Mutation Positive NSCLC (ITT Population) Treated With Erlotinib Plus Tivantinib Compared to Single Agent Chemotherapy.
Description: Progression is defined using Response Evaluation Criteria in Solid Tumors (RECIST v 1.1) criteria as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions or progression of existing non-target lesions are also considered progression.
Time Frame: Date of randomization until disease progression per RECIST (v 1.1) or death from any cause, whichever came first, assessed up to 24 months.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Tivantinib Plus Erlotinib Arm | Chemotherapy Arm
Number analyzed (Participants) | 51 | 45
weeks | 7.3 [6.86 to 24.14] | 18.6 [7.0 to 25.0]
Statistical Analysis 1: Comparison: Tivantinib Plus Erlotinib Arm vs Chemotherapy Arm; Test type: Superiority; p = 0.5017, Log Rank

2. Secondary Outcome: Overall Survival (OS) Among All Eligible Subjects (ITT Population) Treated With Erlotinib Plus Tivantinib Compared to Chemotherapy.
Description: OS is calculated from the date of randomization until death from any cause.
Time Frame: Date of randomization to the date of death from any cause, assessed up to 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tivantinib Plus Erlotinib Arm | Chemotherapy Arm
Number analyzed (Participants) | 51 | 45
months | 6.8 [4.97 to 10.70] | 8.5 [6.37 to 13.97]
Statistical Analysis 1: Comparison: Tivantinib Plus Erlotinib Arm vs Chemotherapy Arm; Test type: Superiority; p = 0.4356, Log Rank

3. Secondary Outcome: Objective Response Rate (ORR) Among All Eligible Subjects (ITT Population) Treated With Erlotinib Plus Tivantinib Compared to Chemotherapy.
Description: Per RECIST v1.1, Complete Response (CR) = disappearance of all lesions and Partial Response (PR) = at least 30% decrease in the sum of diameters of target lesions. ORR = (CR+PR)/# subjects.
Time Frame: Date of randomization to the date of death from any cause or to the date that the subject discontinues from the study, assessed up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Tivantinib Plus Erlotinib Arm | Chemotherapy Arm
Number analyzed (Participants) | 51 | 45
Participants | 0 | 4

4. Secondary Outcome: ORR Among Subjects in the Crossover Period Treated With Erlotinib Plus Tivantinib
Description: Per RECIST v1.1, CR = disappearance of all lesions and PR = at least 30% decrease in the sum of diameters of target lesions. ORR = (CR+PR)/# subjects.
Time Frame: as for outcome 3
Measure: Count of Participants; unit: Participants
Groups:
- Tivantinib Plus Erlotinib Crossover Period: Following radiographically-confirmed progression, subjects randomly assigned to receive chemotherapy had the option to receive erlotinib plus tivantinib and were followed for post-progression objective response rate. Subjects who elected to crossover followed the Erlotinib plus Tivantinib Arm Schedule of Visits, following a post-chemotherapy 21-day washout period, until discontinuation criteria were met.
Arm/Group | Tivantinib Plus Erlotinib Crossover Period
Number analyzed (Participants) | 26
Participants | 2

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the date of the first dose of study drug and up to 30 days after the last dose of study medication.
Arm/Group | Tivantinib Plus Erlotinib Arm | Chemotherapy Arm
All-Cause Mortality (participants affected / at risk) | 3/51 | 4/45
Serious Adverse Events (participants affected / at risk) | 19/51 | 25/45
Other Adverse Events (participants affected / at risk) | 51/51 | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tivantinib Plus Erlotinib Arm (N=51) | Chemotherapy Arm (N=45)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 4
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Aortic valve incompetence (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Disease progression (General disorders) | 3 | 4
Fatigue (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Bacteraemia (Infections and infestations) | 2 | 1
Endocarditis (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 4
Sepsis (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 0 | 2
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to oesophagus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Embolic stroke (Nervous system disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Embolism (Vascular disorders) | 2 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tivantinib Plus Erlotinib Arm (N=51) | Chemotherapy Arm (N=45)
Anaemia (Blood and lymphatic system disorders) | 22 | 22
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 7
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 4 | 7
Neutropenia (Blood and lymphatic system disorders) | 3 | 16
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 9
Arrhythmia (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Cardiomegaly (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 3 | 2
Pericardial effusion (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 2 | 4
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Hyperacusis (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 1
Dry eye (Eye disorders) | 0 | 1
Eye pain (Eye disorders) | 1 | 0
Lacrimation increased (Eye disorders) | 2 | 4
Ocular discomfort (Eye disorders) | 0 | 2
Photopsia (Eye disorders) | 0 | 2
Vision blurred (Eye disorders) | 1 | 2
Vitreous floaters (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Abdominal tenderness (Gastrointestinal disorders) | 1 | 1
Cheilitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 14 | 11
Diarrhoea (Gastrointestinal disorders) | 22 | 14
Dry mouth (Gastrointestinal disorders) | 4 | 1
Dyspepsia (Gastrointestinal disorders) | 5 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 3
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Lip disorder (Gastrointestinal disorders) | 1 | 0
Lip swelling (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 17 | 21
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1
Paraesthesia oral (Gastrointestinal disorders) | 0 | 1
Retching (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 1
Tongue discolouration (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 8 | 8
Asthenia (General disorders) | 3 | 3
Catheter site erythema (General disorders) | 1 | 0
Catheter site pain (General disorders) | 0 | 1
Chest discomfort (General disorders) | 3 | 4
Chest pain (General disorders) | 5 | 3
Chills (General disorders) | 0 | 3
Face oedema (General disorders) | 0 | 2
Facial pain (General disorders) | 2 | 0
Fatigue (General disorders) | 23 | 26
Feeling of body temperature change (General disorders) | 1 | 0
Gait disturbance (General disorders) | 1 | 1
Generalised oedema (General disorders) | 0 | 1
Influenza like illness (General disorders) | 0 | 1
Injection site pain (General disorders) | 0 | 1
Injection site swelling (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 3 | 2
Nodule (General disorders) | 0 | 1
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 6 | 11
Pain (General disorders) | 1 | 2
Pyrexia (General disorders) | 2 | 8
Swelling (General disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Temperature intolerance (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 0
Bronchitis (Infections and infestations) | 1 | 2
Cellulitis (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 1 | 0
Genital herpes (Infections and infestations) | 0 | 1
Herpes virus infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 2
Influenza (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 1
Nasopharyngitis (Infections and infestations) | 0 | 2
Oral candidiasis (Infections and infestations) | 1 | 4
Oral herpes (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 6 | 3
Rash pustular (Infections and infestations) | 2 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Sialoadenitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 2 | 1
Tooth infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 2
Urinary tract infection (Infections and infestations) | 3 | 7
Vaginal infection (Infections and infestations) | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1
Wound abscess (Infections and infestations) | 1 | 0
Contrast media reaction (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 2
Alanine aminotransferase increased (Investigations) | 4 | 4
Aspartate aminotransferase increased (Investigations) | 2 | 3
Blood alkaline phosphatase decreased (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 2
Blood bilirubin increased (Investigations) | 5 | 1
Blood chloride decreased (Investigations) | 1 | 1
Blood creatinine increased (Investigations) | 3 | 5
Blood lactate dehydrogenase increased (Investigations) | 2 | 3
Blood phosphorus decreased (Investigations) | 1 | 0
Blood phosphorus increased (Investigations) | 0 | 1
Blood urea increased (Investigations) | 0 | 1
Brain natriuretic peptide increased (Investigations) | 1 | 0
Breath sounds abnormal (Investigations) | 1 | 0
CD4 lymphocytes decreased (Investigations) | 1 | 0
Fibrin D dimer increased (Investigations) | 0 | 1
Haematocrit decreased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 2 | 1
Neutrophil count decreased (Investigations) | 1 | 2
Neutrophil count increased (Investigations) | 0 | 1
Orthostatic heart rate response increased (Investigations) | 0 | 1
Protein total decreased (Investigations) | 2 | 0
Transaminases increased (Investigations) | 3 | 1
Troponin I increased (Investigations) | 0 | 1
Urine output decreased (Investigations) | 0 | 1
Weight decreased (Investigations) | 6 | 3
White blood cell count decreased (Investigations) | 2 | 2
White blood cell count increased (Investigations) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 17 | 16
Dehydration (Metabolism and nutrition disorders) | 0 | 4
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 9
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 7 | 6
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 8
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 6 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 7
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Haemangioma of bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ageusia (Nervous system disorders) | 0 | 1
Aphasia (Nervous system disorders) | 0 | 1
Brain oedema (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 3 | 6
Dysarthria (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 6 | 5
Dysgraphia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 5
Hyperaesthesia (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 1
Memory impairment (Nervous system disorders) | 1 | 0
Migraine with aura (Nervous system disorders) | 0 | 1
Motor dysfunction (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 2 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 5
Paraesthesia (Nervous system disorders) | 1 | 1
Restless legs syndrome (Nervous system disorders) | 2 | 0
Sciatica (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 2
Syncope (Nervous system disorders) | 1 | 1
Tremor (Nervous system disorders) | 1 | 2
Vasogenic cerebral oedema (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 6 | 9
Confusional state (Psychiatric disorders) | 1 | 2
Delirium (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 5 | 6
Insomnia (Psychiatric disorders) | 3 | 8
Mental status changes (Psychiatric disorders) | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 2
Incontinence (Renal and urinary disorders) | 1 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 2
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Oliguria (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 2 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Breast discomfort (Reproductive system and breast disorders) | 0 | 1
Breast mass (Reproductive system and breast disorders) | 0 | 1
Penile erythema (Reproductive system and breast disorders) | 1 | 0
Varicocele (Reproductive system and breast disorders) | 1 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 10
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 14
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 8
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 14 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 3 | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 3
Nail bed disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 0
Rash (Skin and subcutaneous tissue disorders) | 22 | 7
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1
Embolism (Vascular disorders) | 1 | 0
Flushing (Vascular disorders) | 1 | 1
Hot flush (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 3 | 2
Hypotension (Vascular disorders) | 0 | 7
Lymphoedema (Vascular disorders) | 0 | 2
Microangiopathy (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 1
Phlebitis (Vascular disorders) | 0 | 1
Phlebitis superficial (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No